CLINICAL TRIAL: NCT02558686
Title: Effects of Eccentric Exercise, Sham or Placebo on Post-Needling Soreness by Dry Needling on Active Trigger Points
Brief Title: Exercise and Post-dry Needling Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Head Division, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URJC 2015-12
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Shoulder Pain
Keywords: trigger points; disability; post-dry needling soreness; eccentric exercise
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Eccentric Exercise (Experimental): Individuals will perform 3 sets of 10 repetitions of eccentric exercise of the infraspinatus muscle after the application of trigger point dry needling
  Interventions: Other: Eccentric Exercise
- Detuned Ultrasound (Sham Comparator): Individuals will received 10 minutes of detuned ultrasound on the infraspinatus muscle after the application of trigger point dry needling
  Interventions: Other: Detuned Ultrasound
- Placebo (Placebo Comparator): Individuals will not perform any action after the application of trigger point dry needling
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Eccentric Exercise — Individuals will perform 3 sets of 10 repetitions of eccentric exercise of the infraspinatus muscle after the application of trigger point dry needling
  Arms: Eccentric Exercise
Other: Detuned Ultrasound — Individuals will received 10 minutes of detuned ultrasound on the infraspinatus muscle after the application of trigger point dry needling
  Arms: Detuned Ultrasound
Other: Placebo — Individuals will not perform any action after the application of trigger point dry needling
  Arms: Placebo

SUMMARY:
Application of trigger point dry needling can induce post-dry needling soreness. This is not a negative experience, but sometimes some patients want to reduce it as much as possible. Manual therapies and exercise strategies targeting to decrease post-dry needling soreness need to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral non-traumatic shoulder pain
* Shoulder pain from at least 6 months
* Shoulder pain of more than 3 points on a NPRS
* Presence of active trigger point in the infraspinatus muscle

Exclusion Criteria:

* bilateral shoulder pain
* younger than 18 or older than 65 years
* shoulder injury
* upper extremity surgery
* fibromyalgia syndrome
* neck or shoulder surgery
* cervical radiculopathy
* whiplash
* any type of intervention for the neck-shoulder the previous year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in post-dry needling pain intensity before and after the intervention | Baseline, 24 hours after, 48 hours after and 72 hours after treatment
  A Numerical Pain Rate Scale (NPRS, 0-10) will be used to record post-dry needling soreness and pain

SECONDARY OUTCOMES:
Changes in spontaneous shoulder pain before and after the intervention | Baseline and 72 hours after treatment
  A Numerical Pain Rate Scale (NPRS, 0-10) will be used to assess spontaneous shoulder pain
Changes in disability before and after the intervention | Baseline and 72 hours after treatment
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire will be used to assess disability induced by shoulder pain.
Changes in functionality before and after the intervention | Baseline and 72 hours after treatment
  The Shoulder Pain and Disability Index (SPADI) questionnaire will be used to assess function of the uppr extremity related to shoulder pain

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Fernández-de-las-Peñas, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain